CLINICAL TRIAL: NCT02149693
Title: Paradigm Shift in Medical Education: Applications of High-Fidelity Simulation, Teamwork Model Development, and Concept of Flipped Classroom in Innovation and Revolution of Resuscitation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201401065RIND
Record Dates: First submitted 2014-05-25; First posted 2014-05-29 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2018-12

CONDITIONS: Skill Acquisition of Resuscitation
Keywords: Flipped classroom; High-fidelity simulation; Medical education reform; Medical teamwork; Resuscitation training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- high-fidelity simulation and teamwork training (Experimental): high-fidelity simulation and teamwork training
  Interventions: Other: high-fidelity simulation and teamwork training
- traditional resuscitation training (Active Comparator): traditional resuscitation training
  Interventions: Other: traditional resuscitation training

INTERVENTIONS:
Other: high-fidelity simulation and teamwork training
  Arms: high-fidelity simulation and teamwork training
Other: traditional resuscitation training
  Arms: traditional resuscitation training

SUMMARY:
Medical education was transformed from mainly didactic class before 19th century to the clerkship and internship training based on the concept of "learning by doing" in 20th century. There are new challenges for medical education in the 21th century, including knowledge explosion, the importance of communication and teamwork in clinical care, and lack of comprehensive and systemic experiential learning. Therefore, another paradigm shift of medical education in this century is necessary. This research project, through applying high-fidelity simulation, resuscitation teamwork model, and concept of flipped classroom in resuscitation training, take the innovation and reform of resuscitation training as a pilot test for paradigm shift of medical education.

This research project is a 4-year project. Three innovative intervention for resuscitation training will be developed, implemented, and evaluated. There will be 4 phases in this project:

1. Development phase (1st year): establishment of structure, validity and reliability test, faculty development, and course preparation.
2. Experiment phase (2nd year): comparative studies will be conducted.
3. Implementation phase (3rd year): integration and implementation of innovative interventions.
4. Evaluation phase (4th year): effectiveness evaluation and analysis of learning retention.

Through innovation, development, implementation and effectiveness evaluation in this 4 phases, this research project hope to integrate high-fidelity simulation, resuscitation teamwork model, and concept of flipped classroom, into resuscitation training successfully and appropriately. Furthermore, these experiences can provide the bases of paradigm shift in medical education in the future.

ELIGIBILITY:
Inclusion Criteria:

Health care workers in the following department of National Taiwan University Hospital ward. The Department of surgery, the Department of internal medicine, the Department of Emergency Medicine, the Department of Ambulatory Service.

Exclusion Criteria:

Physical conditions are unsuitable for personnel to implement emergency skills training.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-08; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
resuscitation skill performance | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Wei Yang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan